CLINICAL TRIAL: NCT01865474
Title: DLBS1033 Therapy in Improving Hypercoagulation State in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of DLBS1033 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033-0212
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DLBS1033, Type 2 DM, fibrinolytic, hypercoagulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Thrombophilia | interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment I (Experimental): DLBS1033 bioactive fraction tablet 490 mg thrice daily
  Interventions: Drug: DLBS1033
- Treatment II (Experimental): Placebo tablet of DLBS1033, thrice daily
  Interventions: Drug: placebo tablet of DLBS1033

INTERVENTIONS:
Drug: DLBS1033 — 1 DLBS1033 tablet 490 mg thrice daily for 2 months
  Other Names: Disolf
  Arms: Treatment I
Drug: placebo tablet of DLBS1033 — 1 placebo tablet of DLBS1033 thrice daily for 2 months
  Other Names: placebo tablet of Disolf
  Arms: Treatment II

SUMMARY:
This is a prospective, double-blind, randomized, and controlled study. The investigational product, DLBS1033 at a dose of 490 mg thrice daily or placebo, will be given for an 8-week course of therapy.

DLBS1033 effectively demonstrated fibrinolytic, fibrinogenolytic as well as antithrombotic activities. Hypercoagulation state with high fibrinogen level is usually found in diabetes mellitus patients.

Therefore, the hypothesis of interest of this study is that DLBS1033 will reduce fibrinogen level of diabetes mellitus patients better than that of the Control Group.

DETAILED DESCRIPTION:
There will be 2 groups of treatment, each consisting of 68 subjects, with the treatment regimens as the following:

Treatment I : DLBS1033 bioactive fraction tablet @ 490 mg, three times daily. Treatment II : Placebo tablet of DLBS1033, three times daily.

Clinical examination to evaluate the efficacy of the investigational drug will be performed at baseline and every follow-up visit (at interval of 4 weeks) over the 8 weeks of study period. All subjects will be advised to follow such a lifestyle modification throughout the study period.

All subjects will be under direct supervision of a medical doctor during the study period.

During the study period, anti-diabetes treatment taken by study subjects should still be continued. Other treatment related to subjects' concomitant illnesses, such as hypertension, and/or dyslipidemia, is allowed during subjects' participation in the study.

Other medication such as anti-platelets, fibrinolytic agents and anti-coagulants, or other treatment including herbals/alternatives which may affect haemostatic system, are not allowed to be used during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as type 2 diabetes mellitus with A1c > 7.0% at Screening.
* Men or women, between 25-65 years of age.
* Have been being treated with lifestyle intervention and/or any oral anti-diabetic agents and/or insulin.
* Adequate liver function: ALT and AST ≤ 2.5 times upper limit of normal.
* Adequate renal function: serum creatinine < 2.0 times upper limit of normal.
* Able to take oral medication.

Exclusion Criteria:

1. For females of childbearing potential: Pregnancy, breast-feeding, the intention of becoming pregnant.

   * Patients must accept pregnancy tests during the trial if menstrual cycle is missed.
   * Fertile patients must use a reliable and effective contraceptive.
2. The presence of clinically significant electrocardiographic abnormality
3. History of acute coronary syndrome (myocardial infarction, stroke, unstable angina pectoris), peripheral arterial diseases, venous thromboembolism or other cardiovascular events.
4. History of other arteriosclerotic disease necessitating medical or pharmacological treatment.
5. Severe hypertension (systolic blood pressure ≥ 180 mm Hg, diastolic ≥ 110 mm Hg).
6. Treatment with antiplatelets or antithrombotic agents, including other oral lumbrokinase products within 14 days prior to Screening.
7. Subjects with prior experience with DLBS1033.
8. Subjects with high-risk of bleeding
9. Presence of malignancies as observed clinically or by anamnesis.
10. Subjects with any other disease state, including chronic or acute systemic infections, or uncontrolled illnesses, which judged by the investigator, could interfere with trial participation or trial evaluation.
11. Subjects with known or suspected allergy to study medication or similar products.
12. Subjects with concurrent herbal (alternative) medicines or food supplements suspected to have effect on the primary efficacy endpoint.
13. Subjects enrolled in another experimental (interventional) protocol within the past 30 days prior to Screening.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Fibrinogen level reduction | 8 weeks
  Fibrinogen level reduction from baseline to the end of study (Week 8th)

SECONDARY OUTCOMES:
Change of D-dimer | 4 weeks and 8 weeks
  Change of D-dimer from baseline to every follow-up visit
Change of von Willebrand Factor activity | 4 weeks and 8 weeks
  Change of von Willebrand Factor activity from baseline to every follow-up visit.
Change of hs-CRP level | 4 weeks and 8 weeks
  Change of hs-CRP level from baseline to every follow-up visit.
Change of HbA1c | 8 weeks
  Change of HbA1c from baseline to end of study (Week 8th).
Liver function | 8 weeks
  Liver function (serum ALT, AST,γ-glutamyl transferase, alkaline phosphatase) at baseline and end of study (Week 8th)
Renal function | 8 weeks
  Renal function (serum creatinine, BUN) at baseline and end of study (Week 8th)
Prothrombin Time (PT) | 4 weeks and 8 weeks
  Prothrombin time from baseline to every follow-up visit
Activated partial thromboplastin time (aPTT) | 4 weeks and 8 weeks
  Activated partial thromboplastin time (aPTT)from baseline to every follow-up visit
Adverse events | 4 weeks and 8 weeks (during 8 weeks)
  Adverse events (mainly: GI bleeding, and other bleeding events) from baseline to every follow-up visit
Change of Thromboxane-B2 level | 4 weeks and 8 weeks
  Change of Thromboxane-B2 level from baseline to every follow-up visit (as an indirect indicator to assess the effect of study treatment on TxA2)

CONTACTS AND LOCATIONS:
Overall Officials: Asman Manaf, Prof. Dr. dr., SpPD-KEMD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, University of Andalas/ dr. M. Djamil Padang Hospital, Padang, Sumatera Barat, Indonesia
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, University of Andalas/ dr. M. Djamil Padang Hospital, Padang, West Sumatra, Indonesia